CLINICAL TRIAL: NCT01934205
Title: An Open-label Study To Evaluate Plasma and Pulmonary Pharmacokinetics Following Intravenous Administration of GSK2140944 in Healthy Adult Subjects (BTZ116666)
Brief Title: To Evaluate Plasma and Pulmonary Pharmacokinetics of GSK2140944
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 116666
Record Dates: First submitted 2013-08-29; First posted 2013-09-04 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Infections, Bacterial
Keywords: GSK2140944; pharmacokinetics; bronchoalveolar lavage; pulmonary; antimicrobial; healthy volunteer
MeSH Terms: conditions — Bacterial Infections | interventions — gepotidacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (12):
- Part A(Cohort1) (Experimental): Study BTZ116666 has two parts. Each part will consist of a maximum of 6 cohorts. Part A will be initiated with 4 initial cohorts/timepoints in order to minimize the number of healthy volunteers that undergo bronchoscopy in this study. After review of data from Cohorts 1 through 4 of Part A, the study team will determine if additional cohorts are needed to be studied in Part A and/ or if Part B is needed. If the study team determines that additional cohorts are needed, then only the necessary cohorts in Parts A and/or B will be executed. In Part A, participants will receive GSK2140944 1000 mg intravenous (IV) infusion over 2 hours x 1 dose
  Interventions: Drug: GSK2140944 (Single dose)
- Part A (Cohort2) (Experimental): In Part A, participants will receive GSK2140944 1000 mg intravenous (IV) infusion over 4 hours x 1 dose
  Interventions: Drug: GSK2140944 (Single dose)
- Part A (Cohort3) (Experimental): In Part A, participants will receive GSK2140944 1000 mg intravenous (IV) infusion over 8 hours x 1 dose
  Interventions: Drug: GSK2140944 (Single dose)
- Part A (Cohort4) (Experimental): In Part A, participants will receive GSK2140944 1000 mg intravenous (IV) infusion over 12 hours x 1 dose
  Interventions: Drug: GSK2140944 (Single dose)
- Part A (Cohort5) (Experimental): In Part A, participants will receive GSK2140944 1000 mg intravenous (IV) infusion. Optional Cohort or Part and will only be used if necessary. Sampling times are to be determined based on the review of preliminary PK results from prior study parts and/or cohorts.
  Interventions: Drug: GSK2140944 (Single dose)
- Part A (Cohort6) (Experimental): In Part A, participants will receive GSK2140944 1000 mg intravenous (IV) infusion. Optional Cohort or Part and will only be used if necessary. Sampling times are to be determined based on the review of preliminary PK results from prior study parts and/or cohorts.
  Interventions: Drug: GSK2140944 (Single dose)
- Part B (Cohort1) (Experimental): In Part B, participants will receive GSK2140944 1000 mg IV infusion, q12h x 5 doses. Optional Cohort or Part and will only be used if necessary. Sampling times are to be determined based on the review of preliminary PK results from prior study parts and/or cohorts.
  Interventions: Drug: GSK2140944 (Multiple dose)
- Part B (Cohort2) (Experimental): In Part B, participants will receive GSK2140944 1000 mg IV infusion over, q12h x 5 doses. Optional Cohort or Part and will only be used if necessary. Sampling times are to be determined based on the review of preliminary PK results from prior study parts and/or cohorts.
  Interventions: Drug: GSK2140944 (Multiple dose)
- Part B (Cohort3) (Experimental): In Part B, participants will receive GSK2140944 1000 mg IV infusion over, q12h x 5 doses. Optional Cohort or Part and will only be used if necessary. Sampling times are to be determined based on the review of preliminary PK results from prior study parts and/or cohorts.
  Interventions: Drug: GSK2140944 (Multiple dose)
- Part B (Cohort4) (Experimental): In Part B, participants will receive GSK2140944 1000 mg IV infusion over q12h x 5 doses. Optional Cohort or Part and will only be used if necessary. Sampling times are to be determined based on the review of preliminary PK results from prior study parts and/or cohorts.
  Interventions: Drug: GSK2140944 (Multiple dose)
- Part B (Cohort5) (Experimental): In Part B, participants will receive GSK2140944 1000 mg IV infusion over, q12h x 5 doses. Optional Cohort or Part and will only be used if necessary. Sampling times are to be determined based on the review of preliminary PK results from prior study parts and/or cohorts.
  Interventions: Drug: GSK2140944 (Multiple dose)
- Part B (Cohort6) (Experimental): In Part B, participants will receive GSK2140944 1000 mg IV infusion over, q12h x 5 doses. Optional Cohort or Part and will only be used if necessary. Sampling times are to be determined based on the review of preliminary PK results from prior study parts and/or cohorts.
  Interventions: Drug: GSK2140944 (Multiple dose)

INTERVENTIONS:
Drug: GSK2140944 (Single dose) — A lyophilized formulation, pale yellow to grayish yellow cake containing 750 mg of GSK2140944 (as free base) per vial, Administered intravenously as a single dose.
  Arms: Part A (Cohort2); Part A (Cohort3); Part A (Cohort4); Part A (Cohort5); Part A (Cohort6); Part A(Cohort1)
Drug: GSK2140944 (Multiple dose) — A lyophilized formulation, pale yellow to grayish yellow cake containing 750 mg of GSK2140944 (as free base) per vial, Administered intravenously every 12 hours for 5 doses (3 days).
  Arms: Part B (Cohort1); Part B (Cohort2); Part B (Cohort3); Part B (Cohort4); Part B (Cohort5); Part B (Cohort6)

SUMMARY:
Antimicrobial penetration can be assessed through evaluation of antimicrobial concentrations in various lung compartments, including bronchial mucosal tissue, epithelial lining fluid (ELF), and alveolar macrophages (AM). Antimicrobial concentrations determined in ELF and alveolar macrophages represent an ideal estimate of concentrations at the site of infection and can be accessed via bronchoalveolar lavage (BAL). However sampling of antimicrobial concentrations via BAL is not routine in clinical practice due to its complex methodology and poor patient tolerability. This study will evaluate intrapulmonary and plasma pharmacokinetics of GSK2140944 after single IV dose in adult healthy volunteers. This is a Phase I, open-label study to evaluate plasma and pulmonary pharmacokinetics following intravenous administration of GSK2140944 in healthy adult participants. Part A will evaluate the single dose PK profiles. Part B is optional and will only be conducted if necessary. Each part will consist of a maximum of 6 cohorts. In Part A, only 4 of the 6 cohorts will be dosed initially; cohorts 5 and 6 are optional and will only be dosed if additional time-points are necessary to adequately model the pulmonary pharmacokinetic profile.

ELIGIBILITY:
Inclusion Criteria:

* Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), alkaline phosphatase and bilirubin <=1.5x Upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, vital signs, electrocardiograms (ECGs), physical examination, and laboratory tests. A participant with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included if in the Investigator's judgement the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male or female between 18 and 55 years of age inclusive, at the time of signing the informed consent. A female participant is eligible to participate if she is of non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea. To confirm post-menopausal status, a blood sample for simultaneous follicle stimulating hormone (FSH) > 40 milli-international units per milliliter (MlU/ml) and estradiol < 40 picrograms (pg)/ml (<147 picromoles/Liter [pmol/L]) is confirmatory. Male participant with female partners of child-bearing potential must agree to use one of the contraception methods listed as per protocol. This criterion must be followed from the time of the first dose of study medication until the final follow-up visit.
* Body weight >= 50 kg and Body mass index (BMI) within the range 19 - 31Kilograms/meter^2(kg/m^2) (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* Contraindications to bronchoalveolar lavage including hypercapnia >50 millimeters of mercury (mm Hg), known or suspected intolerability to medications necessary for bronchoscopy, refractory hypoxemia, reactive airway disease or asthma, unstable angina or acute myocardial infarction in the last 6 months, heart failure, and severe hemostatic alterations.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening or positive Human Immunodeficiency Virus (HIV) antibody.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Any clinically significant central nervous system (e.g., seizures), cardiac, pulmonary, metabolic, renal, hepatic or gastrointestinal conditions or history of such conditions that, in the opinion of the investigator may place the participant at an unacceptable risk as a participant in this trial or may interfere with the absorption, distribution, metabolism or excretion of drugs.
* A positive urine test for drugs of abuse or alcohol (or alcohol breath test) at screening.
* A screening urinalysis positive for protein or glucose (greater than "trace" findings of protein or glucose).
* A serum creatinine value that is out of the normal range, or an increase of 0.2 milligrams/decilitre (mg/dL) (or 15.25 micromoles/Liters [µmol/L]) in serum creatinine value between screening and Day -1 visit.
* History of photosensitivity to quinolones.
* Unwillingness to commit to avoid excessive exposure to sunlight (or exposure whilst on a tanning bed) which would cause a sunburn reaction from first dose up to and including the follow-up visit.
* History of drug abuse within 6 months of the study or a history of smoking or use of nicotine containing products within 3 months of screening, or a positive urine cotinine indicative of smoking at screening.
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 grams (g) of alcohol: 12 ounces (360 ml) of beer, 5 ounces (150 ml) of wine or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* The participant has participated in a clinical trial and has received a drug or a new chemical entity within 30 days or 5 half-lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of current study medication.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication, or use of St. John's Wort within 14 days prior to the first dose of study medication. By exception, the volunteer may take paracetamol or acetaminophen (<=2 grams/day) up to 48 hours prior to the first dose of study medication. However, the Investigator and GSK study team can review medication on a case by case basis to determine if its use would compromise participant safety or interfere with the study procedures or data interpretation.
* History of sensitivity to any of the study medications, including GSK2140944 and those that may be used in association with the BAL procedure, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Donation of blood in excess of 500 mL within 12 weeks prior to dosing.
* History of tendon rupture.
* History of sensitivity to heparin or heparin-induced thrombocytopenia (if the clinical research unit uses heparin to maintain intravenous cannula patency).
* Consumption of red wine, pomegranate, seville oranges, grapefruit or grapefruit juice, pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices containing such products from 7 days prior to the first dose of study medication.
* Exclusion criteria for screening ECG (a single repeat is allowed for eligibility determination): Heart Rate, Males <40 and >100 Beat Per Minute (bpm), females <50 and >100 bpm; PR interval <120 and >220 msec; QRS duration <70 and >100 msec; A QT interval corrected for heart rate using the Bazett's formula (QTcB) or Single QT duration corrected for heart rate by Fridericia's formula (QTcF) interval >450 msec. Evidence of previous myocardial infarction (does not include ST segment changes associated with repolarization). A participant has Bundle Branch Block. Any conduction abnormality (including but not specific to left or right complete bundle branch block, AV block [2nd degree or higher], Wolf Parkinson White [WPW] syndrome), sinus pauses>3 seconds, non-sustained or sustained ventricular tachycardia (>=3 consecutive ventricular ectopic beats) or any significant arrhythmia which, in the opinion of the principal investigator and GSK medical monitor, will interfere with the safety of the individual participant.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2013-09-25 (Actual); Primary Completion 2013-12-21 (Actual); Study Completion 2013-12-21 (Actual)

PRIMARY OUTCOMES:
Pulmonary pharmacokinetics of GSK2140944 following intravenous single-dose administration. | Day 1, Day 2, Day 3
  Blood samples will be collected assessment of PK parameters including Epithelial Lining Fluid (ELF) and Alveolar Macrophages (AM) (AUC[0- τ]), Area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration within a participant across all treatments (AUC[0-t]), Maximum observed concentration (Cmax), Time of occurrence of Cmax (tmax), ELF and AM/plasma ratios for GSK2140944 at the early, mid and late dosing interval timepoints, and AUCELF/AUC plasma and AUCAM/AUC plasma ratios, as data permit.
Plasma pharmacokinetics of GSK2140944 following intravenous single-dose administration. | Day 1, Day 2, Day 3
  Blood sample will be collected for estimation of relative bioavailability and assessment of PK parameters including maximum observed concentration; Cmax, area under the concentration-time curve from time 0 to time t; AUC (0-t) and area under the concentration-time curve from time 0 to infinity; AUC(0-infinity), Systemic clearance of parent drug (CL), Volume of distribution at steady state of parent drug after intravascular (e.g., IV) administration (Vdss) and Terminal phase half-life (t½).
Pulmonary pharmacokinetics of GSK2140944 following repeat daily multiple intravenous dose administration. | Day1, Day 2, Day 3, Day 4, Day 5
  Blood samples will be collected assessment of PK parameters including ELF and AM AUC(0- τ)), AUC(0-t), Cmax, tmax, ELF and AM/plasma ratios for GSK2140944 at the early, mid and late dosing interval timepoints, and AUCELF/AUC plasma and AUCAM/AUC plasma ratios, as data permit.
Plasma pharmacokinetics of GSK2140944 following repeat daily multiple intravenous dose administration. | Day1, Day 2, Day 3, Day 4, Day 5
  Blood sample will be collected for estimation of relative bioavailability and assessment of PK parameters including maximum observed concentration; Cmax, area under the concentration-time curve from time 0 to time t; AUC (0-t) and area under the concentration-time curve from time 0 to infinity; AUC(0-infinity), Systemic clearance of parent drug (CL), Volume of distribution at steady state of parent drug after intravascular (e.g., IV) administration (Vdss) and Terminal phase half-life (t½).

SECONDARY OUTCOMES:
Characterisation of the safety profile of GSK2140944 with adverse events (AEs) following intravenous single-dose administration | Up to study day 15
  AE is defined as Any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Characterisation of the safety profile of GSK2140944 with chemistry and haematology laboratory values following intravenous single-dose administration | Up to study day 15
  Any abnormal laboratory test results (haematology, clinical chemistry, or urinalysis)
Characterisation of the safety profile of GSK140944 electrocardiograms (ECG) following intravenous single-dose administration | Up to study day 15
  Twelve (12)-lead ECGs will be obtained using an ECG machine that automatically calculates heart rate and measures PR, QRS, QT, RR and QTcB intervals.
Characterisation of the safety profile of GSK2140944 with vital signs following intravenous single-dose administration | Up to study day 15
  Vital sign measurements will include systolic and diastolic blood pressure, body temperature, pulse rate.
Characterisation of the safety profile of GSK2140944 with adverse events (AEs) following repeat daily multiple intravenous dose administration | Up to study day 18
  AE is defined as Any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Characterisation of the safety profile of GSK2140944 with chemistry and haematology laboratory values following repeat daily multiple intravenous dose administration | Up to study day 18
  Any abnormal laboratory test results (haematology, clinical chemistry, or urinalysis)
Characterisation of the safety profile of GSK140944 electrocardiograms (ECG) following repeat daily multiple intravenous dose administration | Up to study day 18
  Twelve (12)-lead ECGs will be obtained using an ECG machine that automatically calculates heart rate and measures PR, QRS, QT, RR and QTcB intervals.
Characterisation of the safety profile of GSK2140944 with vital signs following repeat daily multiple intravenous dose administration | Up to study day 18
  Vital sign measurements will include systolic and diastolic blood pressure, body temperature, pulse rate.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 116666 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/116666?search=study&search_terms=116666#rs
- Available data/document: Annotated Case Report Form: 116666 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116666 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116666 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116666 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116666 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116666 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116666 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register